CLINICAL TRIAL: NCT02929199
Title: Evaluation of Bio Compatibility of Bio-HPP Crown Veneered With Visio.Lign Compared to Lithium Disilicate (E-max) Crown Veneered With E-max Veneering System in Anterior Esthetic Zone (Randomized Clinical Trial)
Brief Title: Effect of Different Types Crowns on Bio Compatibility and Biological Tissue Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Ali Mraweh, assistant lecturer,Fixed Prosthodontic department,MTI University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-218
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-03

CONDITIONS: Personal Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Pressable E- max, an all ceramic crown
  Interventions: Other: All ceramic crown
- Group B (Experimental): BIO-Hpp hybrid crown
  Interventions: Other: Hybrid crown

INTERVENTIONS:
Other: All ceramic crown — Pressed E-Max coping veneered with E-max veneering system
  Other Names: Prosthetic crown
  Arms: group A
Other: Hybrid crown — pressed Bio HPP veneered with Visio-Lign Veneering system
  Other Names: Prosthetic crown
  Arms: Group B

SUMMARY:
The aim of this study compare soft tissue reaction (bleeding, gingival color and texture), bacteria type and count in the gingival sulcus around the restoration margin and sulcus depth of Bio-compatible High performance polymer( Bio-Hpp) restorations to E-max regardless its popularity in the dental field.

DETAILED DESCRIPTION:
Roles and responsibilities:

1. Esra'a Mohamed Ali Mraweh (E.M):Operator, data enterer and corresponding author;Assistant lecturer, Fixed Prosthodontics Department, Modern Technology and Information University (MTI University), Egypt.
2. Dr. Hesham Alansary ( H.A):Main supervisor, data monitoring, auditing Professor, Fixed prosthodontics department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.
3. Nora Helmy (N.H):Outcome assessors and data collection;Assistant Lecturers, Fixed Prosthodontics department, Faculty of Oral and Dental Medicine, Modern Technology and Information University (MTI university), Egypt.
4. Noha Moustafa (N.M):Base line data collection, recruitment, sequence generation, allocation concealment, patient retention and taking participants' consents;Resident, Fixed Prosthodontics Department, Faculty of Oral and Dental Medicine, Modern Technology and Information University (MTI University), Egypt.
5. Eman Desouky (E.D.):Sample size calculation; Statistician,Faculty of Oral and Dental Medicine, Cairo University, Egypt.
6. Evidence Based Dentistry Committee (CEBD): Help in reporting study protocol following SPIRIT guidelines;Faculty of Oral and Dental Medicine, Cairo University, Egypt.
7. Research Ethics Committee (CREC): Protocol reviewer of the clinical trial in order to protect the right, safety, dignity and well-being of the participants.

Faculty of Oral and Dental Medicine, Cairo University, Egypt.

8. Research Plan Committee (CRPC): For ensuring that this clinical trial following the department research plan; Fixed Prosthodontic Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt.

1. Intervention:E.M. will record the crevice depth and bacterial count prior to preparation. E.M. will perform full coverage conservative tooth preparation following principles of all ceramic crown preparation with shoulder sub-gingival finish line of thickness 1mm using tapered stone with flat end attached to high speed headpiece with air and water coolant after local anesthesia has been given as required.After tooth preparation, E.M will take an adequate 2ry Impression using non aqueous Elastomeric impression materials Impregum™F( medium consistency,3M ESPE) and bite registration, Pink Soft wax(Star dental supply)will be taken. E.M will fabricate the temporary restoration using composite resin temporary material Protemp™4 Temporisation Material (3M ESPE) and cemented using non Eugenol Zinc Oxide temporary cement TempBond™ Temporization( Kerr Dental).

   E.M will deliver pressed Bio-compatible High performance polymer (Bio-HPP) frame work veneered with visio.lign system (Bredent) cemented by a self adhesive resin cement
2. Comparator: E.M. will record the crevice depth and bacterial count prior to preparation. E.M. will perform full coverage conservative tooth preparation following principles of all ceramic crown preparation with shoulder sub-gingival finish line of thickness 1mm using tapered stone with flat end attached to high speed headpiece with air and water coolant after local anesthesia has been given as required.After tooth preparation, E.M will take an adequate 2ry Impression using non aqueous Elastomeric impression materials Impregum™F( medium consistency,3M ESPE) and bite registration, Pink Soft wax(Star dental supply)will be taken. E.M will fabricate the temporary restoration using composite resin temporary material Protemp™4 Temporisation Material (3M ESPE) and cemented using non Eugenol Zinc Oxide temporary cement TempBond™ Temporization( Kerr Dental).

   E.M. will deliver Pres-sable E-max (IPS e.max®) framework will be veneered with e-max veneering system (Ivoclar Vivadent) .The finished crown will be cemented by Self-Adhesive resin Cemen taccording to manufacturer instructions.
3. Outcome:(i)Patient satisfaction (bio-compatibility) measure patient satisfaction using data in questionnaire (presence or absence of bleeding.) The main and standard deviation for the questionnaire of patient at the time crown cementation, 3, 6,9 and 12 months will be recorded.

(ii) Clinical biological outcome:

* measure the Crevice depth using periodontal probe and record the depth in millimeters collected a swap from the teeth and Bacterial count will be measured using culture number of cells per millimeter
* The main and standard deviation for all collected data ,at the time of crown cementation, 3, 6,9 and 12 months will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of patients will be 20-40 years old, able to read and sign the informed consent document.
2. Patient will be able to physically and psychologically to tolerate conventional restorative procedures.
3. Patients have no active periodontal or pulpal diseases, no pockets, bone defects or resorption, have teeth with good restorations.
4. Patients with good Occlusion no para-functional habits
5. Patient with teeth with problems indicated for full coverage restoration (e.g. mild to moderate dislocation, coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
6. Patients are willing to return for follow-up examination and evaluation.
7. Patient with sound contralateral tooth to the selected tooth required for full coverage.
8. Patient with root canal treated tooth requiring full coverage restoration

Exclusion Criteria:

1. Patient in the growth stage with partially erupted teeth.
2. Patient with poor oral hygiene and motivation.
3. Patients with periodontal disease, bony defects.
4. Pregnant women's.
5. Patient with psychiatric problems or unrealistic expectations.
6. Patients have no opposing occluding dentition in the area intended for restoration.
7. Patients with MalOcclusion and Parafunctional habits.
8. smokers

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
change in patient satisfaction(bleeding) | 3,6,9 and 12 months
  presence or absence of bleeding is noted in questionnaire.

SECONDARY OUTCOMES:
Clinical biological outcome(crevice depth) | before preparation, immediately after crown delivery, 3, 6, 9 and 12 months
  Crevice depth(mm): measured using Periodontal probe and recorded in millimeters(mm).
Clinical biological outcome(Bacteria count) | before preparation, immediately after crown delivery, 3, 6, 9 and 12 months
  Bacterial account: from the culture specimens, the number of bacteria Cells per millimeter was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Alansary, Professor, Principal Investigator — affiliated; Ahmed Nagiub, Professor, Principal Investigator — Affiliated; Maha Taymour, associate Professor, Principal Investigator — affliliated
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No